CLINICAL TRIAL: NCT03594097
Title: Use of Coconut Nourish and Queen Garnet Plum to Improve Health in an Elderly Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the study sponsor's request to prematurely terminate this study, the numbers of participants enrolled in the study discontinued or some discontinued earlier due to a screening failure.
Sponsor: University of Manitoba (Other)
Collaborators: University of Southern Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HS21905 (B2018:052)
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2021-04

CONDITIONS: Healthy Ageing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment cookies (Experimental)
  Interventions: Other: Treatment cookies
- Control cookies (Active Comparator)
  Interventions: Other: Control cookies

INTERVENTIONS:
Other: Treatment cookies — Plain flour, Coconut Nourish, Queen Garnet Plum, Unsalted Butter, Artificial Sweetener
  Arms: Treatment cookies
Other: Control cookies — Plain flour, Coconut Powder, Unsalted Butter, Artificial Sweetener, Food Colour
  Arms: Control cookies

SUMMARY:
The purpose of this study is to identify whether the combination of coconut Nourish and Queen Garnet plum are able to attenuate ageing-related complications, including muscle mass loss and inflammation. The study endpoints will measure muscle mass as the primary endpoint with blood lipids, glucose, blood pressure, and inflammatory markers serving as some of the secondary endpoints. As the two products are rich in dietary fibre and anthocyanins, respectively, the study outcome will help to understand role of these dietary components in improving complications that are seen quite frequently in elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years and above
* Able to give written informed consent
* Able to read, write and speak English
* Body mass index less than or equal to 30 kg/m^2
* Either do not suffer from a chronic disease or, if suffering from a chronic disease, then key parameters (blood pressure, blood lipids concentration and blood glucose concentrations) are within the normal physiological range
* Either take no chronic medication or have been treated with a stable dosage of medication for at least 3 months as confirmed by family physician.
* Either take no supplements, or have been utilizing supplements in a stable and consistent dose for at least 3 months, and plan to continue taking a stable and consistent dose throughout the entire study.

Exclusion Criteria:

* Smokers
* Consumption of more than 2 alcoholic drinks/day, or > 14 alcoholic beverages a week, or history of alcoholism or drug dependence
* Uncontrolled hypertension, recent stroke or myocardial infarction, hypothyroidism, diabetes mellitus or kidney disease
* Major disability or disorder requiring continuous medical attention and treatment such as chronic heart failure, liver disease, renal failure or cancer, chronic infections or major surgery within 6 months prior to randomization
* Despite taking medication, do not have values for key parameters (blood pressure, blood lipids concentration and blood glucose concentrations) within normal physiological ranges
* Fasting glucose ≥ 5.6 mmol/L
* Triglycerides ≥ 1.7 mmol/L
* Systolic and diastolic blood pressures ≥130/85 mmHg
* High-density lipoprotein cholesterol ≤1.0 mmol/L
* Have gained or lost >10 lbs in the previous 3 months, or plan to lose weight at any time during the study
* History of allergy to coconut, plum, plain flour, butter or milk
* Any planned surgeries during the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Lean mass | 8 weeks
  Measured using dual-energy x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Body weight | 8 weeks
Body mass index | 8 weeks
  Weight and height will be combined to report BMI in kg/m^2
Waist circumference | 8 weeks
Arm circumference | 8 weeks
Wrist circumference | 8 weeks
Calf circumference | 8 weeks
Triceps skinfold | 8 weeks
Five times chair standing test | 8 weeks
Handgrip dynamometer | 8 weeks
Blood pressure | 8 weeks
  Systolic and diastolic pressure will be assessed
Heart rate | 8 weeks
Bone mineral density | 8 weeks
  Measured using DXA
Bone mineral content | 8 weeks
  Measured using DXA
Fat mass | 8 weeks
  Measured using DXA
Blood total cholesterol | 8 weeks
Blood low-density lipoprotein cholesterol | 8 weeks
Blood high-density lipoprotein cholesterol | 8 weeks
Blood triglycerides | 8 weeks
Blood glucose | 8 weeks
Blood C-reactive protein | 8 weeks
Blood interleukin 1 beta | 8 weeks
Blood tumor necrosis factor alpha | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jones, PhD, Principal Investigator — University of Manitoba
Locations (2):
- University of Southern Queensland, Toowoomba, Queensland, Australia
- Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba, Canada